CLINICAL TRIAL: NCT00772434
Title: Assessment of Bleeding Symptoms in Normal Individuals Using a Comprehensive History Phenotyping Instrument
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: AMA-0637
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Bleeding Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A wide variety of individuals are at risk for bleeding, but even though bleeding symptoms are common it is difficult to compare different people's symptoms. Recent research has found that carefully designed surveys can be used to calculate a bleeding score that is useful for diagnosing bleeding disorders, but normal individuals have not been specifically studied in large numbers with a comprehensive survey. Whether factors like race, ethnicity, age, sex, aspirin use, and previous trauma and surgery influence bleeding scores is also unknown. The primary goal of this study is to use a comprehensive computerized questionnaire to record the bleeding symptoms of normal individuals and then assess the range and severity of bleeding symptoms in this normal population.

Secondary goals include determining whether race, ethnicity, age, sex, aspirin use, and previous trauma and surgery correlate with bleeding symptoms.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Self-assessed as being generally healthy.
* Self-assessed as being able to accurately read and answer questions in English about their past medical histories.

Exclusion Criteria:

* A diagnosis of any disorder of hemostasis.
* A diagnosis of any condition associated with an increased risk of bleeding, namely, any current or previous diagnosis of liver or kidney disease, and malignancy requiring treatment within the past year.
* Use of heparin, low-molecular weight heparins, warfarin, clopidogrel, or other medications with known anticoagulant or anti-platelet properties in the past 30 days.
* History, physical, or known laboratory findings suggestive of any other medical or psychological condition that would impair the participant's ability to accurately respond to questions about bleeding symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a variety of community venues including the existing Rockefeller healthy volunteer database, the Tri-Institutional campus, area universities and medical centers, local colleges, and local business bulletin boards.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Answers to bleeding history questions posed in the questionnaire and cofactors, such as participants' age, sex, history of prior hemostatic challenge, ASA use, ethnicity, and race. | During study visit

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Mauer, MD, Principal Investigator — Rockfeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States